CLINICAL TRIAL: NCT05006261
Title: A Mobile Tai Chi Platform for Fall Prevention in Older Adults - Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020P002974
Record Dates: First submitted 2021-07-27; First posted 2021-08-16 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Healthy Aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tele-Tai Chi (Experimental): Tele-Tai Chi intervention
  Interventions: Device: Tele-Tai Chi

INTERVENTIONS:
Device: Tele-Tai Chi — 12-week simplified TC program using the Tele-TC platform at home, with recommended training sessions at least three times a week, and two or more supplementary live sessions.

SUMMARY:
This is a single-arm longitudinal feasibility study for older adults that involves a 12-week home-based Tai Chi program and includes four remote and/or in-person data collection visits. The investigators will collect additional clinical data in a subset of participants who agree to undergo additional assessments in the Motion Analysis Laboratory at the Spaulding Rehabilitation Hospital in Boston, MA during two in-person data collection sessions. The investigators will assess feasibility and acceptability of the Tele-Tai Chi intervention; explore changes in clinically relevant outcome measures including: physical activity, self-efficacy, quality of life, balance, and gait; and evaluate longitudinal changes in Tai Chi proficiency.

DETAILED DESCRIPTION:
The overall goal of the study is to test the delivery of a novel Tele-Tai Chi (TC) intervention in a single-arm feasibility study for community-dwelling TC-naïve older adults. The investigators will assess feasibility and acceptability of the Tele-TC intervention and its specific components through both qualitative and quantitative feedback, as well as the systematic tracking of adherence data to inform future trials and potential clinical use of the Tele-TC system. The investigators will also explore changes in outcome measures including physical activity, self-efficacy, quality of life, and gait, and evaluate changes in TC proficiency.

Over the course of the 12-week program, participants will be assessed 4 times (baseline, two follow-up assessments at 4 and 8 weeks respectively, and a final assessment at 12 weeks).

Study volunteers will be instructed to train on their own at least three times a week and to participate in 1:1 live sessions with TC instructors two or more times during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 60 and 85 years old
* TC naïve (i.e., never practiced TC)
* Self-reported ability to walk continuously for 15 minutes without an assistive device
* Working email address
* Prior experience with and current access to a computer, smart phone or tablet device

Exclusion Criteria:

* Chronic neuromuscular conditions (e.g. Parkinson's disease, multiple sclerosis, stroke)
* Acute medical conditions requiring hospitalization within the past 6 months or that could interfere with the ability of prospective volunteers to safely participate in the study
* Active cancer
* Significant musculoskeletal conditions requiring chronic use of pain medication
* Cognitive impairment (Diagnosed with dementia (self-reported), or Montreal Cognitive Assessment (MoCA)-Blind score < 18)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tele-Tai Chi
Started | 27
Completed | 26
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: years] | 70 [65 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Protocol Adherence
Description: The percentage of Tai Chi home practice sessions completed by participants.
Time Frame: Post-intervention (approximately 12 weeks)
Population: All dataset was considered
Measure: Mean (Standard Deviation); unit: percentage of session completed
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 26
percentage of session completed | 76.81 (37.32)

2. Primary Outcome: Retention
Description: The percentage of participants who complete the study.
Time Frame: Through study completion, approximately 12 weeks from the beginning of the study
Measure: Number; unit: percentage of subject retained
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 26
percentage of subject retained | 100

3. Primary Outcome: System Usability Scale
Description: The scale is based on a 10-item questionnaire with five response options (from Strongly agree to Strongly disagree) in which participants rate the usability of the system. The scale ranges from 0 to 100, with higher scores indicating greater usability.
Time Frame: Post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 24
score on a scale | 87.18 (13.31)

4. Other Pre Specified Outcome: Ease of Use of the Tele-Tai Chi Platform (Qualitative Interview)
Description: Qualitative interview about ease of use of the Tele-Tai Chi platform. The outcome will be the percentage of participants who provide positive feedback regarding the platform's ease of use.
Time Frame: Post-intervention (approximately 12 weeks)
Population: All dataset analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 26
percentage of participants | 85

5. Other Pre Specified Outcome: Changes From Baseline in Activities-specific Balance Confidence (ABC) Scores
Description: Activities-specific Balance Confidence (ABC): 16-item self-report measure in which participants rate their balance confidence to perform motor activities. The minimum score is 0. The maximum score is 100. Positive changes (i.e., higher scores post-intervention) would represent a positive outcome.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete and extreme outliers were eliminated. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 24
score on a scale | 1.48 (33.59)

6. Other Pre Specified Outcome: Changes From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) 29 Scores
Description: The PROMIS 29 instrument is a 29-item questionnaire assessing each of the following domains: anxiety, depression, fatigue, physical function, pain interference, pain intensity, sleep disturbance, and ability to participate in social roles and activities. The minimum score is 4 per domain, except for pain intensity for which the minimum score is 0. The maximum score per domain is 20, except for pain intensity for which the maximum score is 10. For the physical function and the ability to participate in social roles and activities domains a high score is indicative of positive outcome. For the anxiety, depression, fatigue, sleep disturbance, pain interference, and pain intensity a low score is indicative of positive outcome.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 19
score on a scale
  Ability to Participate in Social Roles/Activities | -0.31 (2.31)
  Anxiety/Fear | 0.10 (1.68)
  Depression and Sadness | 0.26 (1.33)
  Fatigue | -0.78 (2.19)
  Pain Interference | -0.42 (1.49)
  Physical Function | 0.21 (0.76)
  Sleep Disturbance | -0.57 (2.08)
  Pain Intensity | -0.26 (1.11)

7. Other Pre Specified Outcome: Changes From Baseline in Physical Activity Scale for the Elderly (PASE)
Description: Physical Activity Scale for the Elderly (PASE): self-reported level of physical activity in individuals aged 65 years or older during the previous 7 days. The score accounts for the type of activities performed and the time of performance of each activity. The minimum score is 0. The scale has theoretical maximum value of 864, if subjects spent 24 hours per day over 7 days engaged in vigorous activities. However, as this is not possible, a maximum value of 400 is typically considered as that would correspond to being engage in vigorous activities for 8 hours per day + more moderate activities for 4.5 hours per day.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 19
score on a scale | 27.73 (71.16)

8. Other Pre Specified Outcome: Changes From Baseline in Trail Making Test A/B Scores
Description: Trail Making Test (TMT): Test to assess executive cognitive function. It has two parts: TMT A (number sequence only) considers visual search, and TMT B (alternating numbers and letters) evaluates executive control. The participant is asked to draw a line between 24 circles randomly arranged on a page that have to be linked in consecutive order. The TMT is scored by how long it takes to complete the test.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis. For the analysis of Part A only 24 patients were considered.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 25
seconds
  Part A | -0.24 (7.81)
  Part B | -3.37 (35.06)

9. Other Pre Specified Outcome: Changes From Baseline in Self-Efficacy Exercise (SEE) Questionnaire
Description: Exercise Self-efficacy Questionnaire (SEE): 9-item questionnaire that focuses on the self-efficacy expectations for exercise for older adults. The minimum score is 0. The maximum score is 90. Positive changes (i.e., higher scores post-intervention) would represent a positive outcome.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 24
score on a scale | -12.6 (19.92)

10. Other Pre Specified Outcome: Changes From Baseline in Tai Chi Proficiency Scores
Description: Tai Chi experts will use video recordings to score proficiency using a developed instrument to score each of the six Tai Chi movements performed by participants. The minimum score is 6. The maximum score is 30 per Tai Chi exercise. Positive changes (i.e., higher scores post-intervention) would represent a positive outcome. The change in Tai Chi proficiency score ranges from -24 to +24. A change equal to 0 represents no change in proficiency.
Time Frame: Change from Baseline at Post-Intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 22
score on a scale | 6.42 (2.86)

11. Other Pre Specified Outcome: Changes From Baseline in Timed-Up-and-Go
Description: Timed-Up-and-Go: Test to determine fall risk. The participant is asked to stand up from a chair, walk 3 meters, turns 180°, walk 3 meters back, and sits back down with back resting against the chair.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 24
seconds | 0.00 (1.20)

12. Other Pre Specified Outcome: Changes From Baseline in Timed-Up-and-Go Dual Task
Description: Dual task Timed-Up-and-Go test: The participant is asked to stand up from a chair, walk 3 meters, turns 180°, walk 3 meters back, and sits back down with back resting against the chair while counting backwards by three.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 24
seconds | 0.08 (1.78)

13. Other Pre Specified Outcome: Changes From Baseline in Single Leg Stance
Description: Balance on each leg (two trials): The participant is asked to stand on one leg for as long as they can up to a maximum of 30 seconds.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 24
seconds
  Left Leg | 1.75 (7.67)
  Right Leg | 0.73 (10.04)

14. Other Pre Specified Outcome: Changes From Baseline in Sit-to-Stand Performance
Description: Sit-to-Stand Test: The participant is asked to stand up from a chair while keeping their arms crossed across their chest and repeat the task as many times as possible during a period of 30 seconds. A higher count of completed repetitions is considered indicative of improved performance.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset is incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 25
score on a scale | 0.04 (1.56)

15. Other Pre Specified Outcome: Postural Sway and Balance on Both Legs With Feet Shoulder-width Apart
Description: Balance on both legs with feet shoulder-width apart: The participant is asked to stand with feet shoulder-width apart for about 20 seconds. A sensor positioned at the waist is used to track the displacement of the center of mass during the 20 second data collection (for each task). The root mean square (RMS) value of the acceleration data collected using the sensor positioned at the waist is estimated in the antero-posterior (AP) and medio-lateral (ML) directions for the middle 15 seconds of each experiment. Data is gathered at baseline and post-intervention and derived for each condition for a total of 4 variables.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis. The root mean square (RMS) value of the acceleration in the antero-posterior (AP) and medio-lateral (ML) directions at the waist sensor was calculated for middle 15 seconds of each experiment.
Measure: Mean (Standard Deviation); unit: millimeters per second squared
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 21
millimeters per second squared
  AP-Baseline | 60.03 (1.30)
  AP-Post Intervention | 60.73 (0.82)
  ML-Baseline | 60.05 (1.36)
  ML-Post Intervention | 60.48 (0.92)

16. Other Pre Specified Outcome: Postural Sway and Balance on Both Legs With Feet Close to Each Other
Description: Balance on both legs with feet close to each other: The participant is asked to stand with feet as close as possible (without contact between the feet) for about 20 seconds. A sensor positioned at the waist is used to track the displacement of the center of mass during the 20 second data collection (for each task). The root mean square (RMS) value of the acceleration data collected using the sensor positioned at the waist is estimated in the antero-posterior (AP) and medio-lateral (ML) directions for the middle 15 seconds of each experiment. Data is gathered at baseline and post-intervention and derived for a total of 4 variables.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: Data analysis was limited only to subjects who completed in the intervention and completed both baseline and post-intervention assessments. The root mean square (RMS) value of the acceleration in the antero-posterior (AP) and medio-lateral (ML) directions at the waist sensor was calculated for middle 15 seconds of each experiment.
Measure: Mean (Standard Deviation); unit: millimeters per second squared
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 20
millimeters per second squared
  AP - Baseline | 60.14 (1.35)
  AP - Post Intervention | 60.57 (0.57)
  ML - Baseline | 59.93 (1.18)
  ML - Post Intervention | 60.35 (0.65)

17. Other Pre Specified Outcome: Normalized-to-height Stride Length
Description: Study participants will undergo an instrumented gait evaluation. Stride length will be defined as the distance from ipsilateral foot contact to the next ipsilateral foot contact during gait. Normalized-to-height stride length will be derived by computing the stride length using the gait evaluation equipment and dividing such value by the height of the study participant.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset is incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 22
unitless
  Normalized Stride Length - Baseline (unitless) | 0.41 (0.04)
  Normalized Stride Length - Post Intervention (unitless) | 0.41 (0.06)

18. Other Pre Specified Outcome: Stride Time Variability
Description: Study participants will undergo an instrumented gait evaluation. Stride time will be defined as the time interval between two consecutive foot contacts of the same limb. Stride time variability will be computed as the standard deviation of the stride time estimates derived using the gait evaluation equipment.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 22
milliseconds
  Stride Time Variability - Baseline | 10.32 (8.79)
  Stride Time Variability - Discharge | 12.27 (14.70)

19. Other Pre Specified Outcome: Changes From Baseline in Activity Level
Description: Physical activity (e.g. number of steps per day) derived using a wrist-worn activity monitor.
Time Frame: Baseline and end of intervention (approximately 12 weeks)
Population: The dataset was incomplete. Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 9
steps per day | 1044 (2526)

20. Other Pre Specified Outcome: Changes From Baseline in Mini-Balance Evaluation Systems Test (MiniBEST)
Description: MiniBEST Test: Test to assess dynamic balance. It is a 14-item test scored using a three-level ordinal scale. This test will be performed only in individuals who are willing to be tested in the laboratory (as opposed to via a remote visit). The minimum score is 0. The maximum score is 28. Positive changes (i.e., higher scores post-intervention) would represent a positive outcome.
Time Frame: Baseline and end of intervention (approximately 12 weeks)
Population: Data analysis was limited only to subjects who completed both baseline and post-intervention assessments in the laboratory.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 8
score on a scale | 0.5 (1.5)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Tele-Tai Chi
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 14/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-Tai Chi (N=26)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (6) — Reports of back pain, including low back pain. Most cases were pre-existing with flares occurring during the study. Others reported non-study related activities as the cause. No relation to intervention, all cases mild.
Flu-like illness (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Reports of flu-like symptoms during study. All cases self-resolved with supportive care.
Fall (Injury, poisoning and procedural complications) | 3 (4) — Reports of falls during non-study-related activities. No medical care required.
Headache (General disorders) | 1 (1) — Reports of headache during non-study-related activities.
Knee Pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Reports of knee pain in participants with pre-existing knee pain.
Delayed Onset Muscle Soreness (Musculoskeletal and connective tissue disorders) | 4 (6) — Reports of muscle soreness primarily related to non-study-related activities.
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) — Reports of skin irritation related to use of wearable devices.
Dizziness (General disorders) | 3 (3) — Reports of dizziness during non-study-related activities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT05006261/Prot_SAP_000.pdf